CLINICAL TRIAL: NCT01894425
Title: Study of the Role of Infection by Human Papillomavirus (HPV) in the Success Rate of Pregnancies Achieved Via Medically Assisted Procreation
Brief Title: Human Papillomavirus and Rate of Pregnancy Achieved Via Medically Assisted Procreation
Acronym: PAPILLO-PMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2012/SD-01; 2013-A00538-37 (Other: RCB number)
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-04

CONDITIONS: Infertility; Sub-fertility; Papillomavirus Infections
Keywords: Medically assisted procreation; Assisted reproductive technology; Human papilloma virus
MeSH Terms: conditions — Infertility; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples collected (semen and cervical smears) will be sent to the Virology Laboratory of the Hôpital St-Eloi, CHU Montpellier, for analysis. After analysis, the remains of viral DNA will be banked for future studies on the Papilloma Virus.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: The study population consists of couples under care for infertility in the participating centers. Gamete donations are not included. Please see inclusion and exclusion criteria.
  Intervention: HPV screening for women Intervention: HPV screening for men

SUMMARY:
The main objective of this study is to investigate the association between the presence of HPV infection in one or both members of infertile/sub-infertile couples and the outcome of pregnancies obtained by assisted reproduction.

The success of assisted medical procreation is defined as achieving a pregnancy resulting in the birth of a living, viable child.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To study the alterations of sperm present in infertile men according to the presence of HPV in semen.

B. Identify the specific HPV genotypes involved.

C. To study a potential link between HPV and embryonic characteristics (as classified by Giorgetti)

D. To study a potential link between HPV and survival of the conceptus: products of miscarriage or stillbirth, duration of pregnancy, birth weight.

E. To study a potential link between HPV and fetal malformations.

ELIGIBILITY:
Inclusion Criteria:

* Both members of each couple must have given their free and informed consent and signed the consent
* Both members of each couple must be members or beneficiaries of a health insurance plan
* The patient (woman) is available for follow-up after a possible pregnancy
* The patient (woman) is under 43 years of age
* The patient (man) is under 60 years of age
* Couple consulting for infertility services in the participating reproductive medicine centers

Exclusion Criteria:

* One or both members of the couple are involved in another study
* One or both members of the couple are in an exclusion period determined by a previous study
* One or both members of the couple are under judicial protection or under any kind of guardianship
* One or both members of the couple refuse to sign the consent
* It is impossible to correctly inform one or both members of the couple
* The patient (woman) has a contra-indication (or an incompatible combination therapy) for treatment necessary for this study
* The source of sperm is a donor (i.e. it is not possible to obtain a sperm sample from the biological father for use in HPV testing).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of couples under care for infertility in the participating centers. Gamete donations are not included.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10-23 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HPV test for participating women (cervicovaginal sample): positive/negative | baseline (day 0)
HPV test for participating men (sperm sample): positive/negative | baseline (day 0)
Birth of a living, viable child (yes/no) | end of pregnancy (expected maximum of 9 months)
type of medically assisted procreation used | baseline (day 0)

SECONDARY OUTCOMES:
HPV genotypes found | baseline (day 0)
Description of spermogram anomalies | baseline (day 0)
Embryo score according to Giorgetti et al 1995 | Embryo transfer (baseline, day 0)
Blastocyte score according to Gardner & Schoolcraft 1999 | Embryo transfer (baseline, day 0)
Percentage of implantable embryos | Baseline (day 0)
BHCG test | Days 13 to 15 after embryo transfer
  Beta HCG - Human Chorionic Gonadotropin (pregnancy test)
Pregnancy confirmed via ultrasound, yes/no | 5 weeks
Pregnancy confirmed via ultrasound, yes/no | 12 weeks
Spontaneous miscarriage before 3 months, yes/no | 3 months
Spontaneous miscarriage after 3 months, yes/no | end of pregnancy (expected maximum of 9 months)
Spontaneous miscarriage, yes/no | end of pregnancy (expected maximum of 9 months)
Histological and HPV testing on miscarriage samplings | end of pregnancy (expected maximum of 9 months)
Days of gestation | end of pregnancy (expected maximum of 9 months)
Appearance of fetal malformations (yes/no) | end of pregnancy (expected maximum of 9 months)
HPV testing on placenta (positive/negative + genotype) | end of pregnancy (expected maximum of 9 months)
Schieve classification according to weeks of gestation and weight of baby | end of pregnancy (expected maximum of 9 months)
weight of baby at birth / days of gestation (g/day) | end of pregnancy (expected maximum of 9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

IPD SHARING:
Plan to Share IPD: No